CLINICAL TRIAL: NCT07257627
Title: An Open-Label, Randomized, Three-Period Crossover Study Comparing the Pharmacokinetics and Pharmacodynamics of Single-Dose THDB0206 Injection at Different Injection Sites in Healthy Chinese Adults
Brief Title: Comparative PK/PD of Single-Dose THDB0206 at Different Injection Sites
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tonghua Dongbao Pharmaceutical Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: THDB0206L03
Record Dates: First submitted 2025-11-14; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-10

CONDITIONS: Healthy Participants

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- THDB0206 injection-Upper Arm (Experimental)
  Interventions: Drug: THDB0206 injection-Upper arm
- THDB0206 injection-Abdomen (Experimental)
  Interventions: Drug: THDB0206 Injection-Abdomen
- THDB0206 injection-Thigh (Experimental)
  Interventions: Drug: THDB0206 Injection-Thigh

INTERVENTIONS:
Drug: THDB0206 injection-Upper arm — Subjects received a single subcutaneous injection of THDB0206 at a dose of 0.2 U/kg in the upper arm.
  Arms: THDB0206 injection-Upper Arm
Drug: THDB0206 Injection-Abdomen — Subjects received a single subcutaneous injection of THDB0206 at a dose of 0.2 U/kg in the abdomen.
  Arms: THDB0206 injection-Abdomen
Drug: THDB0206 Injection-Thigh — Subjects received a single subcutaneous injection of THDB0206 at a dose of 0.2 U/kg in the thigh.
  Arms: THDB0206 injection-Thigh

SUMMARY:
This open-label, randomized, three-period crossover, 8-hour hyperinsulinemic-euglycemic clamp study will compare the pharmacokinetic and pharmacodynamic profiles of THDB0206 after single subcutaneous administration at different injection sites in healthy Chinese adults.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 and ≤40 years at screening.
2. Body mass index (BMI) ≥18 kg/m² and <25 kg/m² at screening; body weight ≥50 kg for males and ≥45 kg for females at screening.
3. At screening, 75 g oral glucose tolerance test (OGTT): fasting venous plasma glucose <6.1 mmol/L and 2-hour post-load venous plasma glucose <7.8 mmol/L.
4. Glycated hemoglobin (HbA1c) ≤6.1% at screening.

Exclusion Criteria:

1. Known or suspected hypersensitivity to the investigational product or related products, or a history of severe allergies to drugs or foods.
2. Insulin release test at screening considered abnormal with clinical significance in the investigator's judgment.
3. Increased risk of thromboembolism, such as known coagulation disorders, (family) history of thrombosis, or relevant arrhythmias (e.g., paroxysmal atrial fibrillation).
4. In the investigator's judgment, a history of alcohol dependence or drug/chemical substance abuse; or positive results on drug screening/breath alcohol testing at screening; or alcohol consumption exceeding 21 units per week (male subjects) or 14 units per week (female subjects).
5. Subjects who smoked on average more than 5 cigarettes per day within 1 year prior to screening and are unwilling to abstain from smoking during the study.
6. Donation of blood or plasma within the past month, or donation of more than 300 mL of blood within 3 months prior to screening.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2024-04-17 (Actual); Primary Completion 2024-12-02 (Actual); Study Completion 2024-12-02 (Actual)

PRIMARY OUTCOMES:
AUCLisp(0-inf) | From 0 to 8 hours
  Area under the insulin lispro plasma concentration-time curve from zero to infinity

SECONDARY OUTCOMES:
Cmax (Lisp) | From 0 to 8 hours
  The maximum plasma concentration of insulin lispro observed
AUCLisp | From 0 to 8 hours
  Area under the insulin lispro plasma concentration-time curve
tmax(Lisp) | From 0 to 8 hours
  Time to reach the maximum insulin lispro plasma concentration
t1/2 | From 0 to 8 hours
  Terminal half-life
CL/F | From 0 to 8 hours
  CL/F
Vz/F | From 0 to 8 hours
  Apparent volume of distribution
AUCGIR | From 0 to 8 hours
  Area under the glucose infusion rate-time curve
GIRtot | From 0 to 8 hours
  Total glucose infusion during clamping
GIRmax | From 0 to 8 hours
  Maximum glucose infusion rate
tGIRmax | From 0 to 8 hours
  Time to reach the maximum glucose infusion rate
Number of participants with abnormal clinical laboratory findings (haematology, biochemistry and urinalysis) | From the first drug administration to the follow-up visit (3 to 10 days after the last drug administration)
Number of participants with abnormal 12-lead ECG parameters (PR, QR, QRS intervals and QTc) | From the first drug administration to the follow-up visit (3 to 10 days after the last drug administration)
Number of participants with abnormal vital signs (body temperature, supine blood pressure and pulse rate) | From the first drug administration to the follow-up visit (3 to 10 days after the last drug administration)
Number of participants with abnormal physical examination (general condition, head and five sense organs, neck, chest, abdomen, spine and limbs, nervous system) | From the first drug administration to the follow-up visit (3 to 10 days after the last drug administration)
Number of participants with hypoglycemia events in each treatment arm | From the first drug administration to the follow-up visit (3 to 10 days after the last drug administration)
Number of participants with injection site reactions (spontaneous pain, tenderness, itching, redness, edema, induration/infiltration, and others) | From the first drug administration to the follow-up visit (3 to 10 days after the last drug administration)
Number of participants with AE and SAE | From the first drug administration to the follow-up visit (3 to 10 days after the last drug administration)

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Sichuan, China

IPD SHARING:
Plan to Share IPD: No